CLINICAL TRIAL: NCT06531876
Title: A Study of Dreem 3S to Evaluate Continuous Wake and Sleep Monitoring for the Diagnosis and Treatment Monitoring of Narcolepsy
Brief Title: Efficacy of the Dreem 3S Ambulatory Sleep Monitoring Device for the Evaluation of Narcolepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beacon Biosignals (Industry)
Collaborators: Kaiser Permanente (Other); Stanford University (Other); Intrepid Research (Unknown); Sleep Insights (Industry); Sleep Management Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D3KAH
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Narcolepsy Type 1; Hypersomnia; Sleep Disorder
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: This study incluldes is an observational study of the Dreem 3S as compared to polysomnography in patients with hypersomnia. Arm A (undiagnosed) will include subjects who are being evaluated for a hypersomnia disorder, but do not yet have a diagnosis and are not yet under treatment. Arm B (Narcolepsy Type 1) will recruit subjects with known Narcolepsy Type 1, who will withdraw from their therapy and undergo a 7 night period of longitudinal sleep monitoring with the Dreem 3S device, followed by synchronous recording with polysomnography equipment and the Dreem device (see details).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Suspected Hypersomnia Arm [Arm A] (Experimental): Subjects being evaluated for a hypersomnia condition at participating sleep clinics will be recruited to Arm A. These subjects will not yet have a diagnosis and not yet be on treatment. These subjects will undergo 1 week of at-home ambulatory monitoring with the Dreem Headband, followed by formal in-lab evaluation with gold-standard polysomnography/multiple sleep latency testing while also using the Dreem Headband.
  Interventions: Device: Dreem 3S recording
- Known Narcolepsy Type 1 Arm [Arm B] (Experimental): Subjects with known Narcolepsy Type 1, under treatment at participating sleep clinics, will be recruited to Arm B. These subjects will be asked to withdraw from their Narcolepsy related medication therapy starting on day -7, undergo 1 week of at-home ambulatory monitoring with the Dreem Headband on days 1-7, and then undergo two consecutive nights of in-lab PSG followed by MSLT while synchronously using the Dreem headband.
  Interventions: Device: Dreem 3S recording

INTERVENTIONS:
Device: Dreem 3S recording — Subjects in both Arms A and B will undergo at-home recording with the Dreem 3S EEG Headband to assess sleep. Subjects will undergo in-lab polysomnography and multiple sleep latency testing while also wearing the Dreem 3S EEG headband system. Arm B participants will be asked to withdraw from some or all of their Narcolepsy related medication therapy for roughly 19 days in order to assess the ability of the Dreem Headband System in characterizing sleep disturbances related to Narcolepsy.

SUMMARY:
This study intends to examine the utility of a home-use EEG-based sleep monitor for the diagnosis and evaluation of disorders of excessive sleepiness, specifically the neurological disorder Narcolepsy Type 1.

DETAILED DESCRIPTION:
Diagnosing hypersomnia conditions (including narcolepsy type 1 [NT1], narcolepsy type 2 [NT2], and idiopathic hypersomnia [IH]) and differentiating them from other conditions is often challenging as symptoms including excessive daytime sleepiness, daytime napping, and disturbed nocturnal sleep are nonspecific and current diagnostic tests are limited. Unfortunately, patients with hypersomnia often demonstrate a discrepancy between self-reported sleep duration and quantitative assessment. This complicates both diagnosis and management, as objective sleep assessment is typically not available over multiple periods. A more natural approach would be to monitor sleep and wakefulness serially and with monitoring, including assessment of total sleep time, rapid eye movement (REM) latency, daytime sleep attacks, daytime sleep/nap duration, and consolidated/non-consolidated nocturnal sleep.

This validation study evaluates the ability of Dreem 3S to capture multiple days of continuous sleep and wake measures in subjects with hypersomnia, particularly in NT1. Primary outcomes will include usability of Dreem 3S by patients with hypersomnia, patient compliance with longitudinal data collection using Dreem 3S at-home, and fidelity of sleep staging of Dreem 3S data to synchronously recorded gold-standard nocturnal PSG and MSLT.

Dreem 3S is an FDA cleared class II medical device, under the OLZ/OLV (PSG devices) product codes for home sleep staging in patients with disturbed sleep.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old.
* Patients must be scheduled for an MSLT for a potential diagnosis of hypersomnia (Arm A only).
* Patients are able/willing to consent and willing to undergo the nocturnal PSG, MSLT, and Dreem 3S monitoring described in the protocol.
* (for Known NT1 arm [Arm B] only) Deemed safe to discontinue prohibited medications as per protocol.
* (for Known NT1 arm [Arm B] only) Agree to discontinue driving and operating heavy machinery while untreated for their condition and according to the PI's judgement.

Exclusion Criteria:

* Patients under 18 years old.
* If a patient is taking a wake promoting drug and is unsafe to temporarily reduce or discontinue the drug during the 2 weeks prior to nocturnal PSG and MSLT due to their occupation, need to drive or operate heavy machinery, role as a primary caretaker, medical risk of temporarily discontinuing from drug therapy, or any other reason at the discretion of the subject's treating physician or study physicians/PIs.
* Patients suffering from mental and/or physical disorders that could interfere with the study protocol or the interpretation of the results (exclusion based on clinical judgment).
* Shift workers or patients working unusual hours will be excluded. 5. Patients with a history of stroke or epilepsy.
* Patients with an implanted hypoglossal nerve stimulator or a diagnosis of moderate to severe sleep apnea (Apnea-Hypopnea Index (AHI) 3% >15) not adherent on positive airway pressure therapy (usage 30-day window prior to enrollment date reveals <70% days use at least hours; patients treated with non-PAP treatments will not be eligible).
* Patients who are unable to sign an informed consent form, or unable to have a legal guardian who is able to sign along with the patient's assent.
* Patients who are deemed ineligible by the site PI or treating physician for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Compliance with Dreem 3S | 1 week
  The primary outcome of this study is the ability of subjects with hypersomnia to utilize the Dreem 3S system over multiple nights.
Consensus sleep staging | Days 9-10 (est)
  Positive percent agreement (PPA) for WAKE stage for human adjudicated automated sleep staging from the Dreem 3S data (test method) as compared to consensus human sleep staging of synchronouslly recorded PSG data (reference method).

SECONDARY OUTCOMES:
Usability | Days 1-7
  Subject assessment of usability of the Dreem device, as measured by the System Usability Scale
24-hour usability | Day 7 (est)
  Percent of a 24 hour period during which subjects will be asked to wear and operate the Dreem 3S Headband device during which interpretable data is collected.
Detailed comparison between adjudicated Dreem derived sleep stages and PSG derived sleep stages | Days 9-10 (est)
  Examination of Positive Predictive Agreement (PPA) for REM, N1, N2, N3 when comparing adjudicated labels derived from Dreem 3S recorded EEG and sleep stages from human adjudicated PSG data.
Comparison of Dreem derived hypnogram based sleep metrics with in-lab PSG | Days 9-10 (est)
  Percentage of REM in the first 120 minutes of the night (starting after unambiguous sleep onset) will be compared from human adjudicated Dreem sleep labels and human adjudicated PSG data.
Agreement of Dreem derived sleep stages to PSG derived sleep stages | Days 9-10 (est)
  Cohen's kappa of agreement will be calculated between human adjudicated automated sleep staging of Dreem 3S data and manual consensus sleep staging of PSG data collected during in-lab nocturnal monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Kaiser Permanente
Locations (4):
- United States (4):
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - Stanford University, Redwood City, California
  - Sleep Insights Medical Associates PLLC, Rochester, New York
  - Intrepid Research, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
Identifiable participant data will not be shared. Only deidentified data will be shared (EEG data, and related sleep metrics).